CLINICAL TRIAL: NCT00005037
Title: Temozolomide in the Treatment of Advanced Non-Small Cell Lung Carcinoma: Phase II Evaluation in Previously Treated and Chemo-Naive Patients
Brief Title: Temozolomide in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067626; P30CA006927 (NIH); FCCC-99032; NCI-G00-1712
Record Dates: First submitted 2000-04-06; First posted 2004-03-16 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Temozolomide

ARMS (1):
- Temozolomide (Experimental): Temozolomide capsule once a day for 42 days every 10 weeks.
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide
Drug: Temozolomide — Temozolomide capsule once a day for 42 days every 10 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate to temozolomide in previously treated (closed to accrual 8/01) and chemotherapy-naive patients with advanced non-small cell lung cancer. II. Determine the freedom from progression median, and 1-year and 2-year survival rates in these patients on this regimen.

OUTLINE: Patients are stratified by prior chemotherapy (yes (closed to accrual 8/01) vs no). Patients receive oral temozolomide daily for 42 days. Treatment repeats every 8 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months.

PROJECTED ACCRUAL: Up to 66 patients (33 per stratum (previously treated stratum closed to accrual 8/01)) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage IIIB, IV, or recurrent non-small cell lung cancer for which no curative therapy with surgery, radiation, or combination chemoradiotherapy exists Chemotherapy-naive patients: No prior chemotherapy OR At least 6 months since prior adjuvant, induction, or radiosensitizing chemotherapy OR Previously treated patients (closed to accrual 8/01): No more than one prior chemotherapy regimen for relapsed or metastatic disease AND/OR No more than one prior adjuvant, induction, or radiosensitizing chemotherapy within the past 6 months Measurable or evaluable disease CNS metastases allowed (previously treated metastases cannot be only site of measurable disease) No brain metastases with prior whole body irradiation

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No other active invasive malignancies

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biologic therapy allowed Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Recovered from prior radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2000-01; Primary Completion 2002-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
response rate in both previously treated and untreated patients.

SECONDARY OUTCOMES:
freedom from progression (FFP) median, 1-year and 2-year survival rates in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Waukesha Memorial Hospital, Waukesha, Wisconsin